CLINICAL TRIAL: NCT06779526
Title: Effect of Four-Week Wellness Program on Sleep and Work Engagement in a Healthcare Organization
Brief Title: Effect of Four-Week Wellness Program on Work Engagement Burnout and Sleep in a Healthcare Organization (WEBS)
Acronym: WEBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WellSpan Health (Other)
Responsible Party: Principal Investigator, Jay Thimmapuram, Academic Hospitalist, WellSpan Health
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: [2126338-4]
Record Dates: First submitted 2025-01-11; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Sleep; Burnout; Work Engagement
Keywords: heartfulness; meditation; work enagement; sleep; burnout
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The demographic data that is collected from the participants will never be available for the PI/co-investigators to see. It will be secure in a password-protected file, and at the end of the study, the data will be de-identified prior to data analysis. Any information that will be collected from participants will be done so during the screening/intake process. If the participant decides to leave the study, the work email address along with all the information will be deleted from the file. Steps taken to make the subjects feel at ease with the process include informing them during intake about all the specific steps involved ahead of time, so they know what to expect. With regards to the didactic sessions, it will be conducted in Webinar mode, which will protect the names and privacy of the participants from one another. After that, participants will not know the other people who are participating. The repeat questionnaires that are sent to the participants will be directly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Comprised of receiving an orientation session regarding the study, attending at least once weekly didactic sessions on Zoom and participating in morning and evening meditation for ten to fifteen minutes daily. A weekly, live online session for 4 weeks consists of 30 minutes of didactics, comprising of a 10 minute introductory talk on a module of meditation, followed by 20 minutes of guided meditation. Participants provided with materials such as guided audio clips to independently follow heartfulness practices (meditation, rejuvenation, and bed-time relaxation) for 20 minutes each day for 4 weeks: 10 minutes Heartfulness meditation in the morning and 10 minutes in the evening before sleeping
  Email reminders were sent weekly containing audio recordings for guided meditation sessions. All study activities were virtual.
  Interventions: Other: Heartfulness Meditation
- Control arm (No Intervention): The control group would not be undergoing any intervention.

INTERVENTIONS:
Other: Heartfulness Meditation — Receiving an orientation session regarding the study, attending once weekly didactic sessions on Zoom for Heartfulness Meditation, and participating in morning and evening meditation for ten to fifteen minutes daily either by themselves or along with the trainer.
  Arms: Intervention Arm

SUMMARY:
The goal of this clinical trial is to learn if having a 4-week heartfulness meditation program in a healthcare organization would

1. decrease burnout
2. improve sleep and work engagement.

Researchers will compare : intervention group : participating in 4 weeks of Heartfulness Meditation with control group: receiving no intervention

Responses to the Utrecht Work Engagement Scale (UWES), Bergen Insomnia Scale (BIS) and two burnout questions will be compared between the study groups at the beginning and end of the intervention period.

DETAILED DESCRIPTION:
The study is an 8-week single-center prospective, randomized, crossover study among healthcare workers in the WellSpan Health System. All participants were asked to answer two demographic questions and responses to the Utrecht Work Engagement Scale (UWES), and Bergen Insomnia Scale (BIS), two burnout questions were requested for a baseline. Participants were randomized to two groups. One of the groups would undergo the intervention first, which comprised receiving an orientation session regarding the study, attending at least once weekly didactic sessions on Zoom, and participating in morning and evening meditation for ten to fifteen minutes daily. The duration of the intervention period was four weeks. During this time, the control group would not be undergoing any intervention. After four weeks, both groups completed the original questionnaire again followed by a 2 week washout period. This was followed by a crossover, allowing the second group to undergo the intervention for four weeks. After four weeks, the final survey was sent to all participants again.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 and willing to participate
* Able to understand the English language as the instructions were in English

Exclusion Criteria:

* Not able to understand English language

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Sleep | From intervention to end of intervention at 4 weeks for each group
  The Bergen Insomnia Scale (BIS) was measured prior to enrollment, at the four-week time point after the first half of the study, and at the end of the study period at 8 weeks for both the groups. The BIS contains six questions relating to sleep and tiredness, and it is scaled based on the number of days per week that participants are experiencing symptoms. 0 means no days during the course of a week, and 7 indicates every day of the week.

SECONDARY OUTCOMES:
Work engagement | From intervention to end of intervention at 4 weeks for each group
  THE UWES scale, designed to study work engagement using three scales: vigor, dedication, and absorption was measured prior to the beginning of the study, at the four-week time point after the first half of the study, and at the end of the study period at 8 weeks for both groups. The UWES questionnaire contains 9 questions, and participants are given a scale from 0 to 6, with 0 being never to 6 being always 10.
Burnout | From intervention to end of intervention at 4 weeks for each group
  Two burnout questions were asked, 1. I feel burned out from my work 2. I have become more callous toward people since I took this job . The scale for answering these questions ranged from never to everyday. This was measured prior to the beginning of the study, at the four-week time point after the first half of the study, and at the end of the study period at 8 weeks for both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- WellSpan Health, York, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No